CLINICAL TRIAL: NCT04688528
Title: A Prospective Randomized Phase 2 Study of Dose and Volume De-escalation Radiotherapy With Sentinel Lymph Nodes Mapping for Contralateral Irradiation in Unilaterally Node Positive Head and Neck Squamous Cell Carcinomas (SEMIRAHN)
Brief Title: Dose De-escalation and Sentinel LN Mapping Driven Radiotherapy of Contralateral Neck in Ipsilateral Node Positive HNSCC
Acronym: SEMIRAHN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Stichting tegen Kanker (Other); KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S63909; FAF-C/2018/1266 (Other Grant/Funding Number: Stichting tegen Kanker / Fondation contre le Cancer)
Record Dates: First submitted 2020-12-18; First posted 2020-12-30 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: HNSCC; Dose and Volume de-escalation in radiotherapy; sentinel lymph nodes mapping
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: Unilateral RT (Experimental): If SPECT/CT shows ipsilateral drainage and the tumor does not cross the midline, the subject will automatically be assigned to Arm A, and will receive ipsilateral Radiotherapy with reduced prophylactic dose outside of the macroscopically involved nodes. The contralateral side of the neck will be spared according to the absence of sentinel lymph node drainage.
  Interventions: Radiation: Dose de-escalation and / or Volume de-escalation
- Arm B: Whole level (Experimental): If SPECT/CT shows contralateral drainage, the subject will be randomized between 'Whole level' and 'SLN alone'.
  Arm B 'Whole Level': on the contralateral side of the neck, the whole level(s) containing the draining sentinel lymph node(s) will be irradiated at the reduced prophylactic dose. The ipsilateral side of the neck will be irradiated conform to arm A.
  Interventions: Radiation: Dose de-escalation and / or Volume de-escalation
- Arm C: SLN alone (Experimental): If SPECT/CT shows contralateral drainage, the subject will be randomized between 'Whole level' and 'SLN alone'.
  Arm C 'SLN alone': on the contralateral side of the neck, only the sentinel node(s) will be irradiated at the reduced prophylactic dose. The ipsilateral side of the neck will be irradiated conform to arm A.
  Interventions: Radiation: Dose de-escalation and / or Volume de-escalation

INTERVENTIONS:
Radiation: Dose de-escalation and / or Volume de-escalation — The dose de-escalation and/or volume de-escalation strategy will be individually adapted in function of the draining pattern of sentinel lymph nodes on the contralateral side of the neck.

SUMMARY:
The study involves head and neck squamous cell carcinomas (HNSCC) of the oral cavity, oropharynx, larynx or hypopharynx with positive nodes on only one side of the neck and no distant metastasis treated by primary (chemo)radiotherapy.

The elective node irradiation on the contralateral side is not always mandatory and the dose may be too high. In this study, we evaluate two strategies: the impact of sentinel lymph node mapping to tailor the volumes to irradiate and the dose reduction.

DETAILED DESCRIPTION:
The risk of lymph drainage to the contralateral side of the neck is limited to maximum 50% of the patients. Moreover, the risk of occult metastases lies between 20 and 40%. As a consequence, the rule of irradiating the contralateral neck with a prophylactic intent ("elective nodal irradiation") in nearly all HNSCC patients roughly doubles the irradiated volume and, hence, increases the risk of developing more frequent and more severe acute and late side effects. The use of sentinel lymph node mapping to assess the contralateral side of the neck should help to determine the individual drainage to the contralateral side of the neck and, in case of drainage, determine which nodes need to be irradiated. The ultimate goal is to reduce the volume irradiated at prophylactic dose to decrease the risk of severe late side effects (volume de-escalation strategy). This strategy is proposed based on the recent completion of a similar study led by the coordinating investigator, together with the head and neck team of the CHU-UCL-Namur, in HNSCC patients without macroscopic nodes in the neck and treated with (chemo)radiotherapy. It was shown that sentinel lymph node mapping helped to safely individualize and de-escalate the elective nodal irradiation volume and significantly reduce the risk of severe late side effects. Anyway, it is unknown if the whole sub-region of the neck containing the sentinel lymph node(s) or the node(s) only should be defined as target volume.

Moreover, the dose used nowadays for elective nodal irradiation, i.e. 50 Gy in fractions of 2 Gy or biologically equivalent, dates back from the 70's. Many arguments (a.o. our better capacity to stage the neck with 3D imaging and the use of concomitant chemotherapy in the majority of node-positive HNSCC) are in favour of dose de-escalation. A multicentric randomized study performed in 100 HNSCC recently showed that the elective dose could be reduced to 40 Gy in fractions of 2 Gy or biologically equivalent, helping to reduce the risk of late dysphagia at 6 months post-radiotherapy. Confirmatory studies need to be performed on larger groups of patients.

The primary aim is to evaluate contralateral regional control (cRC) rate at 2 years in head and neck squamous cell carcinomas (HNSCC) of the oral cavity, oropharynx, larynx or hypopharynx with positive nodes on only one side of the neck and no distant metastasis treated by (chemo)radiotherapy applying a dose- and/or volume de-escalation.

ELIGIBILITY:
Inclusion criteria

1. Written informed consent given according to ICH/GCP and national/local regulations must be obtained prior to any screening procedures.
2. World Health Organization (WHO) performance status 0-1.
3. Age ≥ 18 years.
4. Patients with a pathologically proven invasive HNSCC, including oral cavity, oropharynx (independently of HPV status), larynx or hypopharynx.
5. Decision by Multidisciplinary Tumor Board of primary treatment with radical radiotherapy with or without concurrent chemotherapy (according to the local guidelines).
6. Baseline imaging of the neck:

   1. ≤ 2.5 mm slices CT with iodine injection (independently or during the FDG-PET/CT examination IF acquired in normal diagnostic conditions, i.e. arms along the thorax with diagnostic quality);
   2. MRI not mandatory but allowed, performed according to centres guidelines;
   3. FDG-PET/CT.
7. Tumor characteristics:

   1. cT-classification (8th TNM staging): T1(except T1 of glottis)-T4a (or, for p16+ oropharyngeal tumors classified cT4, if criteria are compatible with cT4a-stage of p16- tumors).
   2. cN-classification (8th TNM staging), as assessed by iodine contrasted CT (or MRI) and FDG-PET:

      * i. mandatorily cN0 contralaterally to the primary tumor (or on one side of the neck for midline primary tumors):

        * 1. smallest diameter < 5 mm in retropharyngeal level (VIIa);
        * 2. smallest diameter of Küttner node (level IIa) < 12 mm;
        * 3. smallest diameter < 10 mm or sum of smallest and largest diameters < 17 mm in any other level;
        * 4. no central necrosis ;
        * 5. maximal standardized uptake value (SUVmax) ≤ 2.2;
        * 6. in dubious cases (typically 2.2 < SUVmax < 4.5 and inconclusive CT or MRI), US-guided FNAC may be required to exclude positive node contralaterally.
      * ii. ipsilaterally positive (if any of the above mentioned criteria is met), i.e. cN1, cN2a, cN2b, ipsilateral cN3b; or cN1 for oropharyngeal p16+ tumors.
   3. No distant metastasis.

Exclusion criteria

1. Patient has history of:

   1. radiotherapy or surgery in the neck with potential impact on lymphatic drainage ("violated neck");
   2. cancer in the last five years (excluding skin basal cell carcinoma, in situ cervix carcinoma and T1 of glottis or lip, completely chirurgically resected (R0) without intervention disturbing cervical lymph drainage);
   3. Absolute contra-indication to iodine contrast injection, even after proper cortisone and cetirizine pre-medication.
2. HNSCC from nose, sinuses, oesophagus, salivary glands or nasopharynx.
3. Non-HNSCC histology.
4. Positive contralateral neck by node size or positive US-FNAC in dubious nodes.
5. Synchronous second malignancy.
6. Distant metastasis.
7. Tumor crossing the midline without contralateral mapping after 99mTc-nanocolloïd injection.
8. Tumor too large to be safely injected, as deemed by the surgeon. In case of doubt, contact may always be taken with the national coordinating investigator to discuss the situation and take a final decision.
9. Any psychological disorder or familial, sociological or geographical condition which, in the investigator's opinion, might jeopardise participant's safety or compliance with the protocol.
10. Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method.

Highly effective methods of birth control are defined as those, alone or in combination, that result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly; such as implants, injectables, combined oral contraceptives, some IUDs, true sexual abstinence (i.e. refraining from heterosexual intercourse during the entire period of risk associated with the Trial treatments) or vasectomised partner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Contralateral regional control (cRC) rate at 2 years | From baseline to 2 years after radiotherapy
  The rate of tumor control in the draining nodal regions of the neck.

SECONDARY OUTCOMES:
Questionnaire assessing the quality of life of patients with head and neck cancer | From baseline to every 2 months in the first year and every 3 months in the second year after radiotherapy.
  Measured by the EORTC QLQ-H&N35 questionnaire.
Questionnaire assessing the quality of life of cancer patients. | From baseline to every 2 months in the first year and every 3 months in the second year after radiotherapy.
  Measured by the EORTC QOL-C30 (version3) questionnaire.
Normal tissue complication probability (NTCP) gain estimation | Time from RT up to 2 years after RT.
  Estimation of the difference in risk of complications for xerostomia, dysphagia and hypothyroidism according to validated NTCP models.
Local Control | Time from RT until local progression or death whichever comes first, up to 2 years after RT.
  Loco-regional control (LRC)
Survival | Time from RT until the occurrence of a new tumor or death whichever comes first, up to 2 years after RT.
  Cancer specific survival
Survival | Time from RT until death from any cause
  Overall survival
Radiotherapy induced toxicity | Time from start of RT up to 2 years after RT
  Acute and Late Toxicity Scoring

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Daisne, Prof. Dr., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (10):
- Belgium (10):
  - ZOL, Genk, Limburg
  - Jessa Ziekenhuis, Hasselt, Limburg
  - OLV Aalst, Aalst
  - UCL Saint-Luc, Brussels
  - Institute Jules Bordet, Brussels
  - University Hospital Gent, Ghent
  - Universitaire Ziekenhuizen Leuven, Leuven
  - AZ Sint-Maarten, Mechelen
  - CHU-UCL Namur, Namur
  - AZ Turnhout, Turnhout

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daisne JF, Installe J, Bihin B, Laloux M, Vander Borght T, Mathieu I, Lawson G. SPECT/CT lymphoscintigraphy of sentinel node(s) for superselective prophylactic irradiation of the neck in cN0 head and neck cancer patients: a prospective phase I feasibility study. Radiat Oncol. 2014 May 28;9:121. doi: 10.1186/1748-717X-9-121. PMID 24885222
- [Result] Longton E, Lawson G, Bihin B, Mathieu I, Hanin FX, Deheneffe S, Vander Borght T, Laloux M, Daisne JF. Individualized Prophylactic Neck Irradiation in Patients with cN0 Head and Neck Cancer Based on Sentinel Lymph Node(s) Identification: Definitive Results of a Prospective Phase 1-2 Study. Int J Radiat Oncol Biol Phys. 2020 Jul 15;107(4):652-661. doi: 10.1016/j.ijrobp.2020.03.021. Epub 2020 Apr 12. PMID 32294522